CLINICAL TRIAL: NCT02858271
Title: An Open-Label, Single-Dose, Phase 1 Study to Assess the Absorption, Metabolism, Excretion, and Pharmacokinetics of [14C]-AKB-9778 in Healthy Male Volunteers
Brief Title: Study to Assess the Absorption, Metabolism, Excretion and Pharmacokinetics of [14C]-AKB-9778
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aerpio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKB-9778-CI-3004
Record Dates: First submitted 2016-07-20; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AKB-9778 (Experimental): Single dose of [14C]-radiolabeled subcutaneous (SC) injection of AKB-9778 in the morning of Day 1
  Interventions: Drug: AKB-9778 subcutaneous injection

INTERVENTIONS:
Drug: AKB-9778 subcutaneous injection

SUMMARY:
Open-label, single-dose, Phase 1 study to assess the absorption, metabolism, excretion and pharmacokinetics of [14C]-AKB-9778 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* BMI 18 - 33 kg/m2

Exclusion Criteria:

* Significant cardiovascular, pulmonary, or renal disease

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percent of radioactive dose recovered in urine and feces | 7 days
Concentration of total radioactivity in blood and plasma | 7 days
Cmax of AKB-9778 and any major metabolites identified | 7 days
Tmax of AKB-9778 and any major metabolites identified | 7 days
AUC of AKB-9778 and any major metabolites identified | 7 days
t1/2 of AKB-9778 and any major metabolites identified | 7 days
Elimination rate of AKB-9778 and any major metabolites identified | 7 days

SECONDARY OUTCOMES:
Incidence of adverse events and change in vital signs and laboratory values | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Buch, PhD, Study Chair — Aerpio Therapeutics

IPD SHARING:
Plan to Share IPD: Undecided